CLINICAL TRIAL: NCT06467682
Title: The Role of a Wearables-track Tele-exercising Program on Cognitive Function and Brain Oxygenation in Patients With Obstructive Sleep Apnea
Brief Title: 12-week Tele-exercise Program in Patients With OSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Vasileios T. Stavrou, Principal Investigator, University of Cyprus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EEBK/EP 2023/60; 101034403 (Other Grant/Funding Number: ONISILOS - University of Cyprus - Marie Skłodowska-Curie)
Record Dates: First submitted 2024-04-26; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea; Cognitive Impairment
Keywords: tele-rehabilitation; tele-exercise; brain health
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12-week intervention tele-exercise program (Other): tele-exercise and tele-rehabilitation
  Interventions: Other: tele-exercise

INTERVENTIONS:
Other: tele-exercise — The 12-week tele-exercise program will be performed and supported via the USTEP digital platform, with each patient taking part in 3 training sessions per week with a 60-min duration period per training session. There will be personalized training sessions: i) warm-up and warm-down, ii) aerobic exercise, and iii) strength exercises. All tele-exercise program participants, will use wearable-based tracking to assessment the cardio-oxygenation.

SUMMARY:
Obstructive sleep apnea (OSA) contributes to a number of adverse health effects, particularly on brain health. Chronic sleep disturbances caused by OSA could adversely affect cognitive health. Exercise is recommended as a non-pharmacological intervention for patients who are intolerant to continuous positive airway pressure (CPAP) and has been shown to have beneficial effects on brain health and cognitive function. The aim of this protocol is to investigate the effects of a 12-week tele-exercise program on cognitive function and specific parameters of brain activity, including brain metabolism and oxygenation, in patients with OSA. The project aims to demonstrate the multi-dimensional relationship between exercise, cognition and brain oxygenation/metabolism. Our local ethics committee has approved the study. Our population sample (group A = OSA with cognitive impairment (CI) and tele-exercise; group B = OSA with CI and no tele-exercise; group C = OSA without CI and no tele-exercise) will undergo assessment both before and after a 12-week tele-exercise intervention program. This assessment will include a comprehensive battery of subjective and objective assessment tests. Data will be analysed according to group stratification. We hypothesize a beneficial effect of tele-exercise on sleep and cognitive parameters and we are confident that this study will raise awareness among healthcare professionals of the brain health benefits of exercise in patients with low compliance to CPAP treatment.

DETAILED DESCRIPTION:
Background: Obstructive sleep apnea (OSA) is characterized by repetitive episodes of obstruction of the upper airway during sleep and leads to intermittent hypoxia, sleep fragmentation, hypercapnia and sympathetic hyperactivity which are associated with multiple adverse effects on health, in particular with brain health. Hyperarousability in OSA has a negative impact on sleep in the macro- and micro-architecture and sleep continuity, both of which are important players in neurogenesis, brain plasticity, alertness, and memory formation and consolidation. Thus, chronic sleep changes caused by OSA could negatively affect cognitive health. Both sleep fragmentation and intermittent hypoxia interfere with brain structure and function, increasing their vulnerability to neurodegenerative diseases. The prevalence of OSA is increasing as it is conjoined with obesity and it tends to elude clinicians' attention, as in only 10% of the population the definitive diagnosis can be established. Almost 80% of OSA patients report declining performance at work while 40% of dementia risk is attributable to modifiable risk factors such as physical inactivity.

Exercise offers a wide variety of benefits for the general population as it improves the cardiopulmonary, and metabolic profile. In addition, exercise is recommended as a low-cost, easily administered, and non-pharmacologic intervention, with positive effect on brain health and cognitive function, mainly by improving the sleep architecture, by enhancing the neurovascular oxygenation process and cerebral oxygenation, by reducing sympathetic overactivity and improving vascular function at rest and during exercise or mental stress. Finally, it has been shown that exercise can counteract the many aspects of decline in the brain's environment, such as the reduced blood flow and the lack of important factors (i.e. brain-derived neurotrophic factor-BDNF) that nurture brain neurons and encourage the growth and development of new neurons and synapses.

Therefore, long-term exercise providing the greatest and longest-lasting benefits e.g. increase cerebral neurovascular dynamics as assessed with functional Near-Infrared Spectroscopy (fNIRS) method and the intensity of exercise being related to cognitive functions such as improve memory after 12-week aerobic exercise and exercise with resistances. The effectiveness of different physical activity programs has not been properly established and some studies suggest that supervised versus self-selected programs might have similar results. In addition, the types of exercise programs in patients with sleep disorders have been addressed in literature. However, it has been noted that compliance in supervised programs in particular those lasting several weeks can often be an important limitation of the studies. Tele-exercising could be a key to overcome this important limitation, however, data on tele-exercising seems to be scarce.

Purpose: The main goal of the study is to explore the impact of a 12-week tele-exercising program on the cognitive profile as well as on specific parameters of brain functions, brain metabolism and brain oxygenation in patients with obstructive sleep apnea, thus highlighting the multidimensional relationship between physical exercise, cognition and brain oxygenation/metabolism. We will therefore apply a 12-week, wearable-track, tele-exercise intervention in patients with a Sleep Apnea Syndrome with and without cognitive impairment and compare the groups outcome on cognition and brain metabolism.

The primary aim of this study is to investigate the extent to which tele-exercise improves cognitive functions in patients with OSA.

For this aim, we will compare the cognitive performance at baseline and at 12-weeks follow-up in 3 groups of patients.

1. Patients with OSA without cognitive impairment
2. Patients with cognitive impairment assigned to a 12-week tele-exercising program
3. Patients with cognitive impairment not assigned to a tele-exercising intervention

For the screening of cognitive impairment and the evaluation of cognitive outcome, the following cognitive tests will be performed:

* Attention/orientation, memory, verbal fluency, language and visuospatial abilities at ADDENBROOKE'S COGNITIVE EXAMINATION - ACE-R.
* Outcome: Changes between baseline and follow-up at ACE-R subdomains' scores
* Executive function and rote memory
* Outcome: Score at Trail Making Test A and B (TMT)
* Verbal episodic memory based on subdomains of encoding process and immediate recall, free and cued recall, recognition and delayed recall
* Outcome: Score in a serial verbal learning task, with control of encoding and recall, according to the modified procedure of Grober and Buschke
* Procedural memory:
* Outcome: performance in a variation of the visual-motor skill-learning task the Mirror Tracing Task (MTT)
* Working memory with subdomains the auditory information processing speed, flexibility and working memory span:
* Outcome: performance in the Modified Paced Auditory Serial Addition Test (PASAT) and in a task for "Transformed Auditory Span".

The secondary aims of this study are:

1. To investigate the extent to which tele-exercise has a positive impact on brain oxygenation and metabolism in patients with OSA.

   Outcome: cerebral oxygenation according to fNIRS-based measure levels of oxy-hemoglobin (HbO) and deoxygenated-hemoglobin (deoxy-Hb) For this aim, we will compare cerebral oxygenation values fNIRS- at baseline and following a 12-week follow-up in the, above mentioned, three groups of patients.
2. Investigate the extent to which tele-exercise has a positive impact on sleep architecture in patients with OSA.

For this aim, we will compare polysomnography quantitative and qualitative parameters as well as scores in sleep/wake questionnaires at baseline and at 12 weeks follow-up in the, above mentioned, three groups of patients.

Outcomes: Change in sleep architecture, sleep staging features and respiratory features in PSG between baseline and 12-weeks follow up.

Participants: We will recruit patients with clinical suspicion of OSA from Sleep Outpatient clinics at the Nicosia General Hospital, Cyprus, to undergo in home-based polysomnography study with portable device [1]. We will perform a screening cognitive test (ACE-R) to identify individuals with cognitive impairment. Patients with OSA and cognitive impairment (CI) will be randomized to two groups: with CI that will undergo the tele-exercise program (TEp) (Group A, N=20) and with CI That will not undergo the TEp (Group B, N=20). A third matched group (Group C) of OSA patients without cognitive impairment (N=20) will act as another control group and will undergo the tele-exercise program. A sample size estimation, based on previous studies showed that 20 patients per group would be sufficient to detect differences in our primary outcome. Groups A and C will carry out a tele-exercise program form Unique Safe Tele-Exercise Project platform (https://ustep.gr), on a 12-week duration. All patients which will be enrolled in our study will receive non-CPAP treatment (delayed therapy). Α feasibility study will precede with 10 OSA patients (Apnea-Hypopnea-Index, AHI >15 events/h) and similar characteristics, for a 12-week period of tele-exercising so as to investigate and record data related to exercise adherence, drop-out and compliance. All patients group they will be recommendations for diet focused on body weight loss as percent of body fat (where required) and sleep position to improve their quality of life (scale score).

Data collected: Study-related assessments include: a) standard lung function testing, followed by the diffusing capacity of the lungs for carbon monoxide according to ATS/ERS guidelines, b) physical fitness tests [6-MWT (meters) , handgrip strength test (kg) and 30s Sit-to-Stand (repetitions)], so as to record and assess O2 consumption (mL/min/kg) and muscle strength (kg), c) the perceptual ability and reaction time test (ms), d) prior to physical fitness tests, will answer questionnaires on: quality and patterns of sleep (PSQI), shifting attention and for selective attention (TMT A and Β), Epworth Sleep Scale (ESS), Karolinska Sleepiness Scale (KSS), cognitive impairment OSA risk (MoCA), and work ability (WAI) (scales scores) and e) assessments to record cerebral oxygenation-oxygenated (μmol/L) and deoxygenated hemoglobin (μmol/L) (fNIRS) during physical fitness tests, reaction time and when answering the questionnaires. All the above assessments will be performed at baseline and at follow-up in 3 months.

Interventions program: The 12-week TEp will be performed and supported by the uStep platform, with each patient taking part in 3 training sessions per week with a 60-min duration period per training session. There will be personalized training sessions: a) warm-up and warm-down (5-min respectively) with the mobility exercises and respiratory exercises for upper and lower limbs, b) aerobic exercise (30-min) with continuous outdoor walking (intensity calculation according HRpeak during 6MWT and self-reported feeling of dyspnea and leg fatigue) and c) multi-joint strength exercises (20-min) to improve the strength of upper and lower limbs (intensity calculation according to muscle strength tests). Participants of the tele-exercise program will use wearable-based tracking, during intervention period, to assessment the cardio-oxygenation.

ELIGIBILITY:
Inclusion criteria

* age ≥18-to-≤70 years,
* apnea hypopnea index (AHI) ≥15 events/h,
* no contraindications (e.g. unstable angina during the previous month, myocardial infarction during the previous month, resting heart rate >120 bpm, systolic blood pressure >180 mmHg and diastolic blood pressure >100 mmHg) for 6-minute walk test (6MWT)
* body mass index (BMI) <40 kg/m2
* without daily physical working strain
* without active self-reported symptoms (fatigue and dyspnea)
* without pregnancy for women
* patients with preexistent musculoskeletal disability will be excluded since their condition might impair maximum exercise capacity
* all participants should speak and read Greek

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to investigate the extent to which tele-exercise improves cognitive functions in patients with OSA | Baseline and after 12-week
  Absolute number (scale score) in both the total score and the domains of the MoCA questionnaire (assessing cognitive impairment), individual patient, between baseline and after 12 weeks of intervention.

SECONDARY OUTCOMES:
To investigate the extent to which tele-exercise has a positive impact on brain oxygenation in patients with OSA. | Baseline and after 12-week
  Absolute number (μmol/L) in brain oxygenation (fNIRS method), individual of patient, between baseline and after 12 weeks of intervention.
To investigate the extent to which tele-exercise has a positive impact on brain metabolism in patients with OSA. | Baseline and after 12-week
  Absolute number (μmol/L) in brain metabolism (fNIRS method), individual of patient, between baseline and after 12 weeks of intervention.
Investigate the extent to which tele-exercise has a positive impact on sleep architecture in patients with OSA. | Baseline and after 12-week
  Percentage change for each sleep stage (REM and non-REM), individual of patient, between baseline and after 12 weeks of intervention.
To investigate to what extent tele-exercise has a positive effect on oxygen saturation during sleep in patients with OSA. | Baseline and after 12-week
  Duration (min) of in-nadir oxygen saturation during sleep, individual of patient, between baseline and after 12 weeks of intervention.
To investigate the extent to which tele-exercise has a positive impact on Apnea Hypopnea Index in patients with OSA. | Baseline and after 12-week
  Absolute number of Apnea Hypopnea Index (events/h), individual of patient, between baseline and after 12 weeks of intervention.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stavrou VT, Pitris K, Constantinidou F, Adamide T, Frangopoulos F, Bargiotas P. The impact of a 12-week tele-exercise program on cognitive function and cerebral oxygenation in patients with OSA: randomized controlled trial-protocol study. Front Sports Act Living. 2024 Sep 6;6:1418439. doi: 10.3389/fspor.2024.1418439. eCollection 2024. PMID 39346497